CLINICAL TRIAL: NCT02056730
Title: The Study of Efficacy and Safety of Calcium Sensing Receptor in Chronic Dialysis Patients
Brief Title: The Study of Efficacy and Safety of REGPARA Drug in Dialysis Patients Have High Blood Levels of Parathyroid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDCU COA no.637/2013; IRB383/56 (Other: Chulalongkorn University)
Record Dates: First submitted 2014-01-28; First posted 2014-02-06 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2015-02

CONDITIONS: Hyperparathyroidism, Secondary
Keywords: chronic hemodialysis patients; Hyperparathyroidism; Regpara; FGF 23
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hyperparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regpara (Experimental): calcium sensing receptor agonist
  Interventions: Drug: calcium sensing receptor agonist

INTERVENTIONS:
Drug: calcium sensing receptor agonist — For the Regpara those taking 25 mg per day to get the default dose and the dose is adjusted according to the levels of calcium and parathyroid hormone. By adjusting the dose of 25 mg every 3 weeks for a period of 12 weeks, the drug is between 25-75 mg dose, with a maximum dose of not more than 100 mg per day (weeks 3, 6, 9).
  Other Names: Regpara

SUMMARY:
The dialysis patient of chronic kidney disease and parathyroid hormone levels greater than or equal to 800 Pg per ml were divided into two groups by randomized 1:1, one group to receive medication and a control group that did not receive the medication. By group to receive in those taking 25 mg per day to get the default dose and the dose is adjusted according to the levels of calcium and parathyroid hormone. By adjusting the dose of 25 mg every 3 weeks for a period of 12 weeks, the drug is between 25-75 mg dose , with a maximum dose of not more than 100 mg per day (weeks 3, 6 , 9).

After a follow-up treatment in weeks 12, 24 and 36 with an blood,ultrasound test parathyroid glands , abdominal x-ray side . To evaluate the changes without the drug .Unless the track during treatment the patients with low blood calcium levels over 8.4 mg per dL . No dose adjustment . regpara while if blood calcium levels less than 7.5 mg per deciliter . Must be stop taking medication for patients in the control group will receive standard treatment . Which consisted of dose vitamin D sterol and parathyroid surgery . Unable to control the level of parathyroid hormone with vitamin D sterol.

While participating in the research are not allowed to adjust the amount of vitamin D sterol in the two groups . But the amount of dialysate calcium phosphate binders and can be adjusted as appropriate to healthcare is fine .

DETAILED DESCRIPTION:
The renal impairment is caused FGF-23 resistance to the congestion of phosphate and stimulate the secretion of parathyroid hormone (PTH) from the parathyroid gland causes secondary hyperparathyroidism. They also found that high levels of FGF-23 is also a risk factor of vascular calcification.

The Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD) is a disorder caused by renal impairment cause abnormalities occurring in the body. Can be summarized into three main parts as follows : 1) The disorders of minerals and hormones (laboratory abnormalities) such as hyperphosphatemia, secondary hyperparathyroidism. 2 ) The disorders of bone (bone abnormalities) , formerly known as renal osteodystrophy 3) The vascular calcification which results happened increase the risk of heart disease and stroke (cardiovascular disease) , broken bones (fractures) and death rate (mortality).

The secondary hyperparathyroidism. PTH secretion from parathyroid glands are more than normal and a major cause of the congestion of phosphate , reduced levels of 1,25-dihydroxyvitamin D [1,25 (OH) 2D] in the blood and a decrease in blood calcium levels decreased calcium levels in the blood is low. will result in a calcium (calcium sensing receptor or CaSR) on parathyroid glands make parathyroid cell signaling and increased PTH secretion .

That PTH increased continuously in the long run will cause the destruction of the bone called bone decay know "osteitis fibrosa". Some patients with a bone fracture. Important characteristics of osteitis fibrosa is an increase of bone destruction(osteoclastic bone resorption). In addition, the bone marrow may also be found associated with bone marrow fibrosis which causes anemia and did not respond to erythropoietin.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient have age more equal 18 year on enrollment date. 2. The patient get the dialysis of 3 times per week 3. The parathyroid hormone level greater than or equal to 800 pg per mL during the screening 4.The calcium level in the blood is greater than or equal to 9 mg per dL.

Exclusion Criteria:

1. The patient had parathyroid gland surgery.
2. The patient have a history of seizures within 12 weeks before randomized.
3. The patient is scheduled for surgery the kidney
4. The patient will expected parathyroid gland surgery within 6 months
5. The liver function have abnormalities, including SGOT, SGPT, more than two fold
6. The patient had history received a drug of bisphosphonates group or expected to be received during the study.
7. The patient had a history of cancer. Pregnant women. Lactating women. And with sepsis -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety of Regpara in chronic dialysis patients with high blood levels of parathyroid | Baseline to 36 week
  Regpara those taking 25 mg per day to get the default dose and the dose is adjusted according to the levels of calcium and parathyroid hormone. By adjusted dose of 25 mg every 3 weeks (weeks 3, 6, 9) for a period of 12 weeks, the drug is between 25-75 mg dose, with a maximum dose of not more than 100 mg per day .

SECONDARY OUTCOMES:
Efficacy of the REGPARA in reducing the FGF23 level | baseline - 36 week
  The Regpara those taking 25 mg per day to get the default dose and the dose is adjusted according to the levels of calcium and parathyroid hormone. By adjusted dose of 25 mg every 3 weeks (weeks 3, 6, 9) for a period of 12 weeks, the drug is between 25-75 mg dose, with a maximum dose of not more than 100 mg per day .

CONTACTS AND LOCATIONS:
Overall Officials: Kearkiat Praditpornsilpa, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn Memorial Hospital, Bangkok, Pathumwan, Thailand

REFERENCES:
- [Derived] Susantitaphong P, Vadcharavivad S, Susomboon T, Singhan W, Dumrongpisutikul N, Jakchairoongruang K, Eiam-Ong S, Praditpornsilpa K. The effectiveness of cinacalcet: a randomized, open label study in chronic hemodialysis patients with severe secondary hyperparathyroidism. Ren Fail. 2019 Nov;41(1):326-333. doi: 10.1080/0886022X.2018.1562356. PMID 31014177